CLINICAL TRIAL: NCT04208477
Title: "The Effect of Stellate Ganglion Block on Brain Haemodynamics and the Inflammatory Response in Moderate and Severe Brain Injury"
Brief Title: "The Effect of Stellate Ganglion Block in Severe Brain Injury"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Ivan Kostadinov, asist Ivan Kostadinov, dr.med.EDRA, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCLjubljana Stellate
Record Dates: First submitted 2019-11-21; First posted 2019-12-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury; Brain Inflammation; Cerebral Vasospasm
Keywords: stellate ganglion block; brain hemodynamics; brain inflammatory response
MeSH Terms: conditions — Brain Injuries, Traumatic; Encephalitis; Vasospasm, Intracranial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BSG patients (Experimental)
  Interventions: Procedure: one site blockade of the stellate ganglion

INTERVENTIONS:
Procedure: one site blockade of the stellate ganglion — Ultrasound guided one site blockade of the stellate ganglion.

SUMMARY:
Blood flow through the brain is reduced after brain damage. Secondary brain ischemia caused by hypoxia and hypotension, further increase the susceptibility of the ischemically compromised brain to secondary impairment during this period. In order to determine whether and to what extent blockage of the stellate ganglion (BSG) affects the blood flow to the injured brain, the investigators will measure the variables of brain blood flow before and after BSG using computed tomography angiography (CTA), trans-cranial Doppler ultrasound (TCD), intracranial pressure (ICP) and perfusion computed tomography (PCT) of the brain. At the same time, the investigators would like to evaluate whether and to what extent BSG affects the aseptic inflammatory brain injury response and the biochemical indicators of brain damage in patients with moderate and severe brain injury.

DETAILED DESCRIPTION:
Hypothesis

Stellate ganglion blockade in patients with moderate and severe brain damage:

1. Increases the diameter of the brain arteries and blood flow through the brain
2. Do not interfere with intracranial pressure
3. Reduces aseptic inflammatory reaction of the damaged brains measured by IL-6 and reduces damage of the brain tissue measured by protein S100B (S100B), neuron specific enolase (NSE) and glial fibrillary acidic protein (GFAP).

Study design and method description

The study will include 40 subjects of both sexes (18-70 years old) with moderate and severe head injury who will be treated surgically and/or conservatively at the Intensive Care Center (CIT) of the Department of Anesthesiology and Intensive Care UKC Ljubljana. The study will include patients who underwent computed tomography angiography of the brain (CTA) and received an intra-parenchymal intracranial pressure monitor electrode (ICP) at admission to the UKC Ljubljana Emergency Center or during CIT treatment. After primary conservative or surgical care, the subjects will be transferred for further treatment at CIT. Subjects will be sedated and mechanically ventilated. To maintain target cerabral perfusion pressure (CPP), the investigators will give an infusion of noradrenaline as needed. The study will not include subjects with primary decompression craniectomy and radiological signs of progression of intracranial hematomas, subjects in a barbiturate coma, and subjects with a norepinephrine dose greater than 0.2 mcg/kg/min. The study will not include pregnant women, children, patients with known hypersensitivity to iodine contrast media and local anesthetics, and patients with poor renal function (estimated glomerular filtration below 30ml / min / 1.73m2).

The research will be conducted during patient treatment at CIT. The investigators will begin the investigation after positive positive opinions from the Medical Ethics Commission of the Republic of Slovenia, and obtained written consent form patient's family members or official legal representatives.

The effect of BSG on brain blood flow and the diameter of brain vessels will be evaluated by CTA, PCT, TCD.

BSG will be done during the first week after admission at CIT on the same patient's side of the ICP position. One hour after BSG, control CTA in PCT will be done. TCD od the left and right middle brain artery (ACM) will be performed one hour before and after BSG.

TCD will be used to measure the rate of blood flow through ACM in systole-Vs in diastole-Vd and pulsatility index (PI). The investigators will compare Vs, Vd values and PI before and after BSG.

Possible changes in the diameter of large brain vessels after BSG will be compared between CTA done at the emergency center or during CIT treatment and a control CTA after BSG. For standard diameter measurement sites, the investigators will take the middle third of M1 and the proximal part of the M2 segment of the ACM, the middle third of the A1 and A2 segments of the anterior brain artery (ACA), the P1 segment and the first part of P2 segment of the posterior brain artery (ACP), the terminal part of the interior carotid artery (ACI), the middle third of the intradural part of the vertebral artery and middle third of the basilar artery. Changes in the diameter of the brain vessels will be presented numerically and descriptively.

With PCT-produced color maps beside qualitative evaluation od the possible changes of the brain blood flow on the left and right brain hemisphere after BSG, the investigators will also evaluate changes in regional brain blood volume (rCBV), regional brain blood flow (rCBF), mean transition time (MTT). Outside the contusion regions, the investigators will mark the region of interest (ROI) of 500 mm2 for ACA, ACM and ACP perfusion areas. Siemens SyngoVia software will be used.

PCT and CTA will be done by the helical CT tomogram (Somatom, Siemens, Erlangen, Germany). A 40 ml non-ionic low-osmolar iodine contrast medium, 370 mg/ml iopromide (Ultravist; Bayer HealthCare, Berlin, Germany) will be used. It will be injected at a flow rate of 5 ml/s into a cubital vein. Perfusion imaging will be initiated 7 seconds after the injection of contrast.

Blood samples for the determination of IL6, NSE, S100B in GFAP will be drawn from the right external jugular vein and peripheral artery (radial or femoral artery) one hour before and 1, 6, 12, 24 hours after BSG. The investigators will compare IL6, NSE, S100B, GFAP values in venous blood from right jugular vein before v after BSG. A comparation of the values of IL6, NSE, S100B, GFAP in venous blood from the right internal jugular vein in arterial blood taken from the peripheral artery will be done as well. Blood samples will be sent for analysis to the central laboratory of UKC Ljubljana.

Brain oxygenation will be measured with a non-invasive method on both fronts using Near Infrared Spectroscopy (NIRS). NIRS measurement values will be measured immediately before BSG and within 5, 10, 15, 20, 25 and 30 minutes after BSG.

BSG will be done ipsilaterally to the inserted ICP electrode. BSG will be done under ultrasound control at the C6-C7 level, with a lateral approach with a Stimulplex Ultra 360 5cm needle (B.Brown). A 6-15 MHz high frequency probe will be used. BSG will be done always by the same anesthesiologist. The injection site and the ultrasound probe will be aseptically prepared. The ultrasound probe will be placed transversely to the neck axis at the height of the sixth cervical vertebra. After preliminary verification of the needle tip position over the long cervical muscle and under the prevertebral fascia and after negative aspiration, 8 ml of 0.5% levobupivacaine will be injected. Because het investigator's subjects will be sedated, onset of the BSG will be confirmed 10 minutes after the blockade, by the onset of three signs of Horner's syndrome (ptosis, myosis, enophthalmus, anhydrosis, conjunctival hyperemia): enophthalmus, anhydrosis, conjunctival hyperemia.

ICP in CPP will be continuously measured before and after BSG. The data will be analyzed in graphical display using IBM SPSS Statistics statistical programs, ver. 25 and Microsoft Excel. The variables will be presented as mean values with standard deviation or as median with interquartile range. Using the paired t-test, the investigators will compare the average values of the sample's numerically variables. Significant differences will be defined as p<0,05.

Expected results

When investigating the effect of BSG on the brain circulation and inflammatory response in subjects with moderate and severe brain damage, the investigators expect a significant increase in the diameter of the large brain arteries, and thus a positive effect of BSG on the brain circulation of the injured brain (decreased mean blood transition time, increased blood volume in the brain, and increased blood flow through the brain). The investigators estimate that BSG will not change the intracranial pressure. The investigators expect NIRS values to be significantly higher after the blockade than before the blockade. Due to the positive effects of BSG on the aseptic inflammatory response of non-injured brain, BSG is expected to have the same effect in the injured brain. The investigators also expect BSG will decrease the concentration of biochemical indicators of inflammation and damage to neurons and glia.

ELIGIBILITY:
Inclusion Criteria:

* patients with moderate and severe head injury
* patients who underwent computed tomograply angiography of the brain (CTA) at admission to the UKC Ljubljana Emergency Center or during CIT treatment
* patients with intra-parenchymal intracranial pressure monitor electrode (ICP) installed

Exclusion Criteria:

* patients with primary decompression craniectomy
* radiological signs of progression of intracranial hematomas
* barbiturate coma
* patients with a norepinephrine dose greater than 0.2 mcg/kg/min
* pregnant women
* children
* known hypersensitivity to iodine contrast media and local anesthetics
* poor renal function (estimated glomerular filtration below 30ml / min / 1.73m2).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in diameter of the cerebral arteries | First measurement of the diameter will be done on the CTA made during the first week of hospitalization. Control measurement will be done 1 hour after the BSG.
  Diameters of the cerebral arteries will be measured in millimeters (mm) on the CTA before and after BSG. Measurement of the diameter will be done on standard positions: middle third of M1 segment and upper part of M2 segment of middle cerebral artery, middle third of A1 and A2 segment of anterior cerebral artery, P1 segment and first part of P2 segment of posterior cerebral artery, terminal part of internal carotid artery, middle third of the intradural part of vertebral artery and middle third of basilar artery.

SECONDARY OUTCOMES:
Change of mean transition time (MTT) on perfusion computed tomography. | Indicators will be measured 1 hour after the BSG
  Measurement will be mede with perfusion computed tomography done after one side BSG (left or right, depending of the side of ICP electrode position). Comparation will be made between left and right hemisphere. Measures will be expressed seconds.
Change of regional cerebral blood flow (rCBF) on perfusion computed tomography. | Measurement will be measured 1 hour after the BSG
  Measurement will be mede with perfusion computed tomography done after one side BSG (left or right, depending of the side of ICP electrode position). Comparation will be made between left and right hemisphere. Measures will be expressed ml/100g brain tissue/min.
Change of regional cerebral blood volume (rCBV) on perfusion computed tomography. | Measurement will be measured 1 hour after the BSG
  Measurement will be mede with perfusion computed tomography done after one side BSG (left or right, depending of the side of ICP electrode position). Comparation will be made between left and right hemisphere. Measures will be expressed ml/100g brain tissue.
Change of systolic velocity (sV) on transcranial Doppler ultrasound | Measurement will be made one hour before and one hour after the BSG.
  With transcranial Doppler measurement of systolic velocity (sV) will be made on middle cerebral artery and expressed in cm/s.
Change of diastolic velocity (dV) on transcranial Doppler ultrasound | Measurement will be made one hour before and one hour after the BSG.
  With transcranial Doppler measurement of diastolic velocity (dV) will be made on middle cerebral artery and expressed in cm/s.
Change of pulsatiloty index on transcranial Doppler ultrasound | Measurement will be made one hour before and one hour after the BSG.
  With transcranial Doppler measurement of pulsatility index will be made on middle cerebral artery.
Change of the brain tissue oxygenation. | Measurements will be made before and 5, 10, 15, 20, 25, 30 minutes after the BSG.
  Brain tissue oxygenation will be measured with near infrared spectroscopy (NIRS) on both sides of the head.
Change of the ICP. | Measurement will be done before and every minute in the next 12 hours after the BSG.
  Intracranial pressure will be measured with the intracranial pressure electrode in mmHg.
Change in concentration of plasma interleucin 6 (IL-6). | Blood samples will be taken 1 hour before BSG. Next samples 1, 6, 12, 24 hours after the BSG.
  The investigators will measure plasma interleucin 6 (IL-6) in micrograms/mL. Blood samples will be taken from arterial line and right deep jugular vein.
Change in concentration of plasma protein S100B (S100B). | Blood samples will be taken 1 hour before BSG. Next samples 1, 6, 12, 24 hours after the BSG.
  The investigators will measure plasma protein S100B in mcg/L. Blood samples will be taken from arterial line and right deep jugular vein.
Change in concentration of plasma neuron specific enolase (NSE). | Blood samples will be taken 1 hour before BSG. Next samples 1, 6, 12, 24 hours after the BSG.
  The investigators will measure plasma neuron specific enolase (NSE) in micrograms/L. Blood samples will be taken from arterial line and right deep jugular vein.
Change in concentration of plasma glial fibrillary acidic protein (GFAP). | Blood samples will be taken 1 hour before BSG. Next samples 1, 6, 12, 24 hours after the BSG.
  The investigators will measure plasma glial fibrillary acidic protein (GFAP) in micrograms/L. Blood samples will be taken from arterial line and right deep jugular vein.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivan Kostadinov, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years

REFERENCES:
- [Derived] Kostadinov I, Avsenik J, Osredkar J, Jerin A, Gradisek P. Effect of stellate ganglion block on brain hemodynamics and the inflammatory response in moderate and severe traumatic brain injury: a pilot study. Reg Anesth Pain Med. 2025 Feb 19:rapm-2024-106185. doi: 10.1136/rapm-2024-106185. Online ahead of print. PMID 39971387